CLINICAL TRIAL: NCT03373669
Title: Effect of Extended Dose Intervals on the Immune Response to Oral Cholera Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00008066
Record Dates: First submitted 2017-12-04; First posted 2017-12-14 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Cholera; Vibrio Cholerae Infection
Keywords: oral cholera vaccine; OCV; dose interval
MeSH Terms: conditions — Cholera | interventions — Cholera Vaccines; shanchol

STUDY DESIGN:
Intervention Model Description: This is an open label, randomized, phase 2 clinical trial of the immunogenicity of OCV when the vaccine is administered to participants of three age cohorts (1-4 years, 5-14 years, and >14 years) and in two dose interval groups (DIGs). The subjects in each age cohort will be randomized to a DIG of 2 weeks (DIG-1) or 6 months (DIG-2). A total of 120 subjects will be enrolled and these are equally divided between the different groups (20 per age/dose interval group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shanchol Dose-interval Group 1 (Active Comparator): Participants in Dose-Interval Group 1 (DIG-1) will receive the oral cholera vaccine, Shanchol, according to the manufacturer instructions: in 2 doses at Day 0 and two weeks later (Day 14).
  Interventions: Biological: Oral Cholera Vaccine
- Shanchol Dose-Interval Group 2 (Experimental): Participants in Dose-Interval Group 2 (DIG-2) will receive the Adjusted Dose oral cholera vaccine, Shanchol, with a delayed second dose. The vaccine will be given at Day 0 and six months later.
  Interventions: Biological: Adjusted Dose Oral Cholera Vaccine

INTERVENTIONS:
Biological: Oral Cholera Vaccine — Shanchol is a bivalent (O1 and O139 serotypes) vaccine using a heat-killed classical Inaba strain and a formalin-killed classical Ogawa strain produced by Sanofi. Shanchol requires no oral buffer for administration, is approved for persons greater than 1 year of age, and requires 2 doses at two-week intervals. It became World Health Organization (WHO) prequalified in 2011.
  Other Names: Shanchol
  Arms: Shanchol Dose-interval Group 1
Biological: Adjusted Dose Oral Cholera Vaccine — The Adjusted Dose Oral Cholera Vaccine is given in two doses, with the second dose given at six months, rather than the manufacturer described 2 week interval between first and second dose.
  Other Names: Shanchol delayed dose
  Arms: Shanchol Dose-Interval Group 2

SUMMARY:
Cholera is a life-threatening disease if prompt actions are not taken. The most recent estimates of the global burden of cholera estimate that there are more than 1.3 billion people at risk. Of which, 2.86 million (range: 1.3-4.0 million) will contract cholera and 95,000 (21,000-143,000) will die each year. A safe, effective, and affordable killed whole-cell oral cholera vaccine (OCV) is now being used widely to prevent cholera in areas at risk. This regimen demonstrated 65% efficacy retained for at least 3 years and even up to 5 years in an endemic setting.

The primary aim of this project is to determine changes in the vibriocidal geometric mean titers (GMT) in subjects who receive the second dose of oral cholera vaccine (OCV) at different intervals: 2 weeks, or 6 months following the first dose of vaccine. Secondary aims include a) vibriocidal antibody response rates in subjects who receive OCV at 2 weeks or 6 months following the first dose of vaccine, b) age specific serum vibriocidal GMTs following the second dose among participants given the second dose of OCV at intervals of 2 weeks or 6 months following the first dose of vaccine, c) GMT and antibody response rates of Immunoglobulin A (IgA) and Immunoglobulin G (IgG) anti-lipopolysaccharide (anti-LPS) as measured by ELISA following the second dose among participants given the second dose of OCV at intervals of 2 weeks or 6 months following the first dose of vaccine. Our hypothesis is that the vibriocidal GMT following the second dose, when given after 6 months will not be inferior to the response when the second dose is given according to the standard interval of two weeks.

DETAILED DESCRIPTION:
Cholera is a life-threatening disease if prompt actions are not taken. The most recent estimates of the global burden of cholera estimate that there are more than 1.3 billion people at risk. Of which, 2.86 million (range: 1.3-4.0 million) will contract cholera and 95,000 (21,000-143,000) will die each year. A safe, effective, and affordable killed whole-cell oral cholera vaccine (OCV) is now being used widely to prevent cholera in areas at risk. This regimen demonstrated 65% efficacy retained for at least 3 years and even up to 5 years in an endemic setting.

As described in the package insert, the standard dosing schedule of the OCV is two doses with the second dose given 2 weeks after the first. In several campaigns, it was felt to appropriate to give a single dose to twice as many people and to give the second dose at a later time when this was logistically possible. In fact, modelling of the impact of OCV during an outbreak finds that when the vaccine supply is limited (as it is currently), more cases are prevented if a single dose strategy is used since a single dose can be provided to twice as many people. Even if the efficacy is a bit lower, the number of cases prevented will be higher. Even the individual person in this situation will be better off if more of his neighbors also receive vaccine since he benefits from the herd protection when more people are vaccinated.

A single dose strategy was used during an outbreak in Zambia in 2015-16, but this first dose was then followed up with a second dose after 6 to 8 months. I was also used in Haiti in 2016-17 following the hurricane. While the delayed second dose strategy has been used and will likely continue to be used during outbreaks or during humanitarian crises, there is no feasible way to assess the relative effectiveness against clinical cholera comparing a two-week interval with a delayed second dose strategy.

While clinical effectiveness trials are not feasible, serological responses comparing different dose intervals are possible. One such study found that vibriocidal titers were similar if the second dose was given either 2 week or 4 weeks after the first , but studies have not been done with longer dose intervals, as was used in Zambia and Haiti.

The proposed study will determine if giving the second dose of the OCV using a longer interval will result in a response to the second dose that is not inferior, or perhaps even results in a more prolonged elevated vibriocidal titre. From an immunological standpoint, there could be advantages to a longer dose interval if this resulted in a true booster response which sustained high titre of antibody. While acknowledging that the vibriocidal titer is not an established correlate of protection, it is the best correlate of the immune response following vaccination. It seems logical that a sustained high titer is likely to be more effective. Unfortunately, the clinical trials comparing the 2 week and 4 week interval with Shanchol only examined the serum titers shortly after the dosing (about 2 weeks). Follow-up serum samples were not obtained to discern how these dose intervals compared in terms of duration of elevated serum titres.

Recent studies have found that children <5 years of age are less well protected than older individuals even though their serum antibody response rates (take rates) were similar to the older subjects when the serum was collected about two weeks after the vaccine doses were administered. These immunogenicity studies have not, however, examined antibody titers when blood samples were obtained after a longer time interval. Therefore, it is not known if the antibody titers decline at the same rate as older subjects. It could be that GMT titers are lower or that titers fall more rapidly in the young children, and a different dosing interval could maintain higher titres. To compare antibody responses in different age groups, we plan to stratify groups into age 1-4, 5-14, and 15 years and older.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥1 year, stratified into different age groups
2. Living in the Waya Clinic Catchment Area
3. Good health condition, without clinically significant medical history (by participant or guardian, in case of minor)
4. Not pregnant for female subjects.
5. Available to participate for the study duration, including all planned follow-up visits for up to 9 months from screening.
6. Signed informed consent

Exclusion Criteria:

1. Presence of a significant medical or psychiatric condition (Examples include: Diagnosis and treatment of tuberculosis (TB) or HIV; renal insufficiency; hepatic disease; oral or parenteral medication known to affect the immune function, such as corticosteroids, other immunosuppressant drugs; or behavioural or memory issues)
2. Ever having received oral cholera vaccine.
3. Receipt of an investigational product (within 30 days before vaccination).
4. History of diarrhoea in 7 days prior to first dose of vaccine (defined as ≥3 unformed loose stools in 24 hours).
5. History of chronic diarrhea (lasting for more than 2 weeks in the past 6 months)
6. Current use of laxatives, antacids, or other agents to lower stomach acidity?
7. Planning to become pregnant in the next 2 years.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Vibriocidal GMT | 6 months
  The primary aim of this project is to determine changes in the vibriocidal geometric mean titers (GMT) in subjects who receive the second dose of oral cholera vaccine (OCV) at different intervals: 2 weeks or 6 months following the first dose of vaccine.

SECONDARY OUTCOMES:
Vibriocidal Antibody Response Rates | 2 weeks and 6 months
  vibriocidal antibody response rates in subjects who receive OCV at 2 weeks or 6 months following the first dose of vaccine.
Age specific vibriocidal response | 2 weeks and 6 months
  age specific serum vibriocidal GMTs following the second dose among participants given the second dose of OCV at intervals of 2 weeks or 6 months months following the first dose of vaccine.
IgG ELISA Antibody Response | 2 weeks and 6 months
  GMT and antibody response rates of IgG anti-LPS as measured by ELISA following the second dose among participants given the second dose of OCV at intervals of 2 weeks or 6 months following the first dose of vaccine.
IgA ELISA Antibody Response | 2 weeks and 6 months
  GMT and antibody response rates of IgA anti-LPS as measured by ELISA following the second dose among participants given the second dose of OCV at intervals of 2 weeks or 6 months following the first dose of vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda K Debes, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Center for Infectious Disease Research - Zambia, Lusaka, Zambia

REFERENCES:
- [Background] Ali M, Nelson AR, Lopez AL, Sack DA. Updated global burden of cholera in endemic countries. PLoS Negl Trop Dis. 2015 Jun 4;9(6):e0003832. doi: 10.1371/journal.pntd.0003832. eCollection 2015. PMID 26043000
- [Background] Sridhar S. An affordable cholera vaccine: an important step forward. Lancet. 2009 Nov 14;374(9702):1658-60. doi: 10.1016/S0140-6736(09)61418-5. Epub 2009 Oct 8. No abstract available. PMID 19819005
- [Background] Bi Q, Ferreras E, Pezzoli L, Legros D, Ivers LC, Date K, Qadri F, Digilio L, Sack DA, Ali M, Lessler J, Luquero FJ, Azman AS; Oral Cholera Vaccine Working Group of The Global Task Force on Cholera Control. Protection against cholera from killed whole-cell oral cholera vaccines: a systematic review and meta-analysis. Lancet Infect Dis. 2017 Oct;17(10):1080-1088. doi: 10.1016/S1473-3099(17)30359-6. Epub 2017 Jul 17. PMID 28729167
- [Background] Bhattacharya SK, Sur D, Ali M, Kanungo S, You YA, Manna B, Sah B, Niyogi SK, Park JK, Sarkar B, Puri MK, Kim DR, Deen JL, Holmgren J, Carbis R, Dhingra MS, Donner A, Nair GB, Lopez AL, Wierzba TF, Clemens JD. 5 year efficacy of a bivalent killed whole-cell oral cholera vaccine in Kolkata, India: a cluster-randomised, double-blind, placebo-controlled trial. Lancet Infect Dis. 2013 Dec;13(12):1050-6. doi: 10.1016/S1473-3099(13)70273-1. Epub 2013 Oct 18. PMID 24140390
- [Background] Kanungo S, Desai SN, Nandy RK, Bhattacharya MK, Kim DR, Sinha A, Mahapatra T, Yang JS, Lopez AL, Manna B, Bannerjee B, Ali M, Dhingra MS, Chandra AM, Clemens JD, Sur D, Wierzba TF. Flexibility of oral cholera vaccine dosing-a randomized controlled trial measuring immune responses following alternative vaccination schedules in a cholera hyper-endemic zone. PLoS Negl Trop Dis. 2015 Mar 12;9(3):e0003574. doi: 10.1371/journal.pntd.0003574. eCollection 2015 Mar. PMID 25764513
- [Derived] Mwaba J, Chisenga CC, Xiao S, Ng'ombe H, Banda E, Shea P, Mabula-Bwalya C, Mwila-Kazimbaya K, Laban NM, Alabi P, Chirwa-Chobe M, Simuyandi M, Harris J, Iyer AS, Bosomprah S, Scalzo P, Murt KN, Ram M, Kwenda G, Ali M, Sack DA, Chilengi R, Debes AK. Serum vibriocidal responses when second doses of oral cholera vaccine are delayed 6 months in Zambia. Vaccine. 2021 Jul 22;39(32):4516-4523. doi: 10.1016/j.vaccine.2021.06.034. Epub 2021 Jul 1. PMID 34217572